CLINICAL TRIAL: NCT03569072
Title: High Intensity Functional Image Guided Vmat Lung Evasion
Acronym: HI-FIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREC/18/PMCC/23; U1111-1208-1546 (Registry Identifier: UTN)
Record Dates: First submitted 2018-05-30; First posted 2018-06-26 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Non Small Cell Lung Cancer Stage III
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalated functionally adapted radiation therapy (Experimental): This is a single arm study
  Interventions: Radiation: Functionally adapted, dose escalated VMAT radiotherapy

INTERVENTIONS:
Radiation: Functionally adapted, dose escalated VMAT radiotherapy — Volumetric Modulated Arc Therapy planning and treatment delivery to treat primary and nodal planning target volume with 60 Gy in 30 fractions and a simultaneous integrated boost to the primary tumour to a total dose 69Gy in 30 fractions while avoiding organs at risk including functional lung, heart and oesophagus.

SUMMARY:
This study is being performed to assess the feasibility of adapting radiotherapy plans based on functional lung information and increasing the dose to the primary tumour. This is a single arm interventional pilot study involving 20 patients.

Aims Primary: to assess the feasibility of using ventilation and perfusion positron emission computed tomography (V/Q PET/CT) scans to adapt radiotherapy plans using Volumetric Modulated Arc Therapy (VMAT) to avoid regions of functional lung and deliver a higher dose to the primary tumour Secondary: to assess the incidence of acute and late radiotherapy toxicities, to quantify regional ventilation loss and regional perfusion loss on post treatment V/Q PET/CT, to assess associations of V/Q PET/CT with other functional lung imaging techniques, to assess overall survival, progression free survival and quality of life outcomes.

Participants: 20 patients stage IIIa-c non-small cell lung cancer for curative intent radiotherapy.

Methods: All patients will receive functional lung adapted 60 Gray (Gy) in 30 fractions to the primary and nodal planning target volume with a simultaneous integrated boost to the primary tumour to a total dose 69Gy in 30 fractions.

Expected outcomes: That functionally adapted lung radiotherapy using V/Q PET/CT imaging and VMAT planning is technically feasible.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Written informed consent has been provided.
* Histologically or cytologically confirmed Non-Small Cell Lung Cancer
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 within 2 weeks prior to registration
* Locally advanced disease (stage IIIA, IIIB, IIIC as per American Joint Committee on Cancer AJCC, 8th ed.) as confirmed on staging 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG) PET/CT
* No evidence of metastatic intracranial disease on CT brain with contrast or MRI
* Willing to participate in the full follow up schedule
* Planned for treatment with curative intent

Exclusion Criteria:

* Participant is not able to tolerate supine position on PET/CT bed for the duration of the PET/CT acquisitions, is not cooperative, or needs continuous nursing (e.g. patient from Intensive Care Unit) or is unable to attend full course of follow up visits
* Pregnancy or Breast-feeding
* If history of a prior extra thoracic invasive malignancy (except non-melanomatous skin cancer) must be free from recurrence for a minimum of 3 years at the time of registration
* Prior radiotherapy to the lungs or mediastinum (a history of prior breast radiotherapy is not an exclusion)
* Prior known history of interstitial lung disease * A history of renal impairment or reaction to iodine contrast is not an exclusion criteria, if a patient has medical comorbidities that exclude the use of iodine contrasts, these exploratory investigations can be omitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Treatment will be considered feasible if all of the following criteria is met: Reduction in mean functional lung dose of ≥2%, functional lung volume receiving 20Gy of ≥4%, Mean heart dose is ≤30 Gy and relative heart volume receiving 50 Gy is <25% | 1 year
  To assess the technical feasibility of the delivery of personalised functional lung radiotherapy.

SECONDARY OUTCOMES:
The number of patients with radiation pneumonitis will be assessed and graded using CTCAE v4.03 | 1 year
  To determine the incidence of grade ≥ 2 clinical or radiological pneumonitis after high dose functionally adapted radiotherapy
Quantitative voxel-wise comparison of ventilation PET/CT measures will be contoured using semi-automatic threshold based on the operator's discretion and compared with the pre-treatment ventilation PET/CT. | 3 months and 12 months following completion of radiotherapy
  To quantify regional ventilation loss on post treatment ventilation PET/CT following functionally adapted lung radiotherapy. Measures will use the end-inspiratory and end-expiratory volume for each lung and lobe. Assessed on V PET/CT imaging from baseline to 3 months post treatment and from baseline to 12 months.
Quantitative voxel-wise comparison of perfusion PET/CT measures will be contoured using semi-automatic threshold based on the operator's discretion and compared with the pre-treatment perfusion PET/CT. | 3 months and 12 months following completion of radiotherapy
  To quantify regional perfusion loss on post treatment ventilation PET/CT following functionally adapted lung radiotherapy. Measures will use the end-inspiratory and end-expiratory volume for each lung and lobe. Assessed on Q PET/CT imaging from baseline to 3 months post treatment and from baseline to 12 months
Quantitative voxel-wise comparison of CT Ventilation with Ventilation PET/CT | 3 months and 12 months following completion of radiotherapy
  To assess the associations between ventilation PET/CT with inhale/exhale CT ventilation. This will be compared on imaging at baseline, 3 months post treatment and 12 month post treatment.
Quantitative voxel-wise comparison of dual energy CT (DECT) iodine mapping with Perfusion PET/CT | 3 months and 12 months following completion of radiotherapy
  To assess the associations between perfusion PET/CT with dual energy CT iodine mapping ventilation (DECT iodine mapping is regarded as a surrogate for pulmonary perfusion). This will be compared on imaging at baseline, 3 months post treatment and 12 month post treatment.
The number of patients with Grade ≥ 2 cardiac toxicity will be assessed and graded using CTCAE v4.03. | 3 months and 12 months following completion of radiotherapy
  This will be assessed by pre, 3 and 12 month post treatment transthoracic echocardiograms and ECG investigations.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas W Bucknell, MBBS (hons), Principal Investigator — Peter Mac Callum Cancer Centre
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaudreault M, Korte J, Bucknell N, Jackson P, Sakyanun P, McIntosh L, Woon B, Buteau JP, Hofman MS, Mulcahy T, Kron T, Siva S, Hardcastle N. Comparison of dual-energy CT with positron emission tomography for lung perfusion imaging in patients with non-small cell lung cancer. Phys Med Biol. 2023 Jan 27;68(3). doi: 10.1088/1361-6560/acb198. PMID 36623318
- [Derived] Bucknell N, Hardcastle N, Jackson P, Hofman M, Callahan J, Eu P, Iravani A, Lawrence R, Martin O, Bressel M, Woon B, Blyth B, MacManus M, Byrne K, Steinfort D, Kron T, Hanna G, Ball D, Siva S. Single-arm prospective interventional study assessing feasibility of using gallium-68 ventilation and perfusion PET/CT to avoid functional lung in patients with stage III non-small cell lung cancer. BMJ Open. 2020 Dec 10;10(12):e042465. doi: 10.1136/bmjopen-2020-042465. PMID 33303468